CLINICAL TRIAL: NCT07288983
Title: A Randomized, Double-Blinded, Controlled Trial Comparing the Analgesic Efficacy and Motor-Sparing Properties of the Pericapsular Nerve Group (PENG) Block, Suprainguinal Fascia Iliaca Compartment Block (S-FICB), and Lumbar Erector Spinae Plane Block (L-ESPB) in Patients Undergoing Hip Arthroplasty
Brief Title: PENG Block vs Suprainguinal FICB vs Lumbar ESPB for Analgesia After Hip Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG block (Active Comparator): Participants in this arm will receive a Pericapsular Nerve Group (PENG) block performed under ultrasound guidance. The block will be administered with 20 mL of 0.2% ropivacaine injected lateral to the iliopsoas tendon at the level of the anterior inferior iliac spine and iliopubic eminence. No additional peripheral nerve blocks will be performed. All participants will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- Suprainguinal FICB (Active Comparator): Participants will receive a suprainguinal Fascia Iliaca Compartment Block (S-FICB) performed under ultrasound guidance. A total of 40 mL of 0.2% ropivacaine will be injected in the suprainguinal fascia iliaca plane to achieve spread toward the femoral nerve, lateral femoral cutaneous nerve, and obturator nerve. All participants will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Interventions: Procedure: Suprainguinal Fascia Iliaca Compartment Block (S-FICB)
- Lumbar ESPB (Active Comparator): Participants will receive a lumbar Erector Spinae Plane Block (L-ESPB) performed under ultrasound guidance at the L4 transverse process level. A total of 20 mL of 0.2% ropivacaine will be injected deep to the erector spinae muscle and superficial to the transverse process. No sacral ESPB will be added. All participants will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Interventions: Procedure: Lumbar Erector Spinae Plane Block (L-ESPB)

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — The Pericapsular Nerve Group (PENG) block will be performed under ultrasound guidance using a curvilinear or linear transducer. A 22-gauge echogenic needle will be advanced in-plane toward the fascial plane between the iliopsoas tendon and the pelvic brim at the level of the anterior inferior iliac spine. A total of 20 mL of 0.2% ropivacaine will be injected incrementally with repeated aspiration to avoid intravascular injection. No additional peripheral nerve blocks will be performed. All patients will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Arms: PENG block
Procedure: Suprainguinal Fascia Iliaca Compartment Block (S-FICB) — The suprainguinal fascia iliaca compartment block will be performed under ultrasound guidance using a high-frequency linear probe placed in the sagittal oblique plane above the inguinal ligament. After identifying the fascia iliaca above the iliacus muscle, a 22-gauge echogenic needle will be advanced in-plane into the suprainguinal fascia iliaca space. A total of 30 mL of 0.2% ropivacaine will be injected to achieve cranial spread toward the femoral nerve, lateral femoral cutaneous nerve, and obturator nerve. All patients will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Arms: Suprainguinal FICB
Procedure: Lumbar Erector Spinae Plane Block (L-ESPB) — The lumbar erector spinae plane block will be performed under ultrasound guidance at the L4 transverse process level. A curvilinear or linear ultrasound probe will be used to identify the erector spinae muscle and underlying transverse process. A 22-gauge echogenic needle will be inserted in-plane and advanced to the fascial plane deep to the erector spinae muscle and superficial to the transverse process. A total of 20 mL of 0.2% ropivacaine will be injected incrementally. No sacral ESPB will be added. All patients will receive standardized spinal anesthesia and multimodal postoperative analgesia.
  Arms: Lumbar ESPB

SUMMARY:
This randomized, double-blinded, controlled clinical trial compares three motor-sparing regional anesthesia techniques used for postoperative analgesia in patients undergoing hip arthroplasty: the Pericapsular Nerve Group (PENG) block, the suprainguinal Fascia Iliaca Compartment Block (S-FICB), and the Lumbar Erector Spinae Plane Block (L-ESPB). Although all three techniques are widely used in modern hip surgery, their relative analgesic efficacy, opioid-sparing potential, and impact on early functional recovery have not been directly compared in a single study.

The primary objective is to determine which block provides the most effective postoperative analgesia while preserving motor function and facilitating early mobilization. Secondary objectives include comparisons of opioid consumption, pain scores at rest and during movement, time to first rescue analgesia, block-related adverse events, quadriceps strength, incidence of postoperative nausea and vomiting, and early functional outcomes.

This study aims to identify the optimal motor-sparing regional anesthesia strategy for older adults undergoing hip arthroplasty.

DETAILED DESCRIPTION:
Regional anesthesia plays a key role in modern multimodal analgesia for hip arthroplasty, particularly in older adults who are vulnerable to opioid-related adverse effects and postoperative functional decline. Several motor-sparing nerve block techniques have been developed to improve postoperative pain control while maintaining quadriceps strength and enabling early mobilization. Among them, the Pericapsular Nerve Group (PENG) block, the suprainguinal Fascia Iliaca Compartment Block (S-FICB), and the Lumbar Erector Spinae Plane Block (L-ESPB) are widely used in clinical practice. However, no randomized clinical trial has directly compared these three approaches within a single study population.

The PENG block targets the articular branches of the femoral, obturator, and accessory obturator nerves, providing selective analgesia of the anterior hip capsule with minimal motor involvement. The suprainguinal FICB delivers a higher spread of local anesthetic over the femoral nerve, lateral femoral cutaneous nerve, and variable portions of the obturator nerve, offering broader sensory coverage but with a higher likelihood of quadriceps weakness. The lumbar ESPB is a posterior fascial plane block that may achieve indirect spread toward the lumbar plexus, potentially providing balanced anterior and posterior capsular analgesia while preserving motor function.

This randomized, double-blinded, three-arm controlled trial aims to compare the analgesic effectiveness, opioid-sparing properties, and motor-sparing characteristics of PENG, S-FICB, and L-ESPB in patients undergoing hip arthroplasty. All participants will receive standardized spinal anesthesia and multimodal postoperative analgesia. The study's primary endpoint is the time to first rescue opioid administration. Secondary outcomes include total postoperative opioid consumption, pain scores at rest and during movement, quadriceps muscle strength, block performance time, incidence of postoperative nausea and vomiting, early mobilization parameters, and block-related adverse events.

The results of this trial are expected to clarify the relative benefits and limitations of the three most commonly used motor-sparing regional anesthesia techniques for hip surgery and to guide optimal selection of blocks for enhanced recovery pathways in older adults undergoing hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older scheduled to undergo elective hip arthroplasty under spinal anesthesia.
* Ability to provide written informed consent.
* Ability to understand and reliably use numerical pain assessment tools (NRS 0-10).
* ASA physical status II-III.
* Expected postoperative hospitalization of at least 48 hours to ensure complete data collection.

Exclusion Criteria:

* Inability to provide informed consent due to cognitive impairment, language barrier, or severe hearing/speech limitations.
* Coagulopathy or therapeutic anticoagulation not meeting safety criteria for regional anesthesia.
* Local infection at the planned block site.
* Allergy, hypersensitivity, or contraindication to ropivacaine, local anesthetics, or study medications.
* Pre-existing lower-limb neurological deficits (motor or sensory) affecting outcome assessments.
* Severe spinal deformity or anatomical limitations preventing safe performance of regional blocks.
* Chronic opioid use (defined as >30 mg oral morphine equivalents daily for more than 2 weeks).
* Severe renal failure (eGFR <30 mL/min/1.73m²) or severe hepatic impairment.
* Uncontrolled diabetes mellitus (fasting glucose >300 mg/dL or HbA1c >10%).
* History of local anesthetic systemic toxicity (LAST).
* Participation in another interventional clinical trial within the past 30 days.
* Any condition deemed by investigators to interfere with protocol adherence, safety monitoring, or outcome reliability.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption in the First 48 Hours After Surgery | 0-48 hours postoperatively
  Total cumulative opioid consumption recorded in the first 48 postoperative hours, converted to morphine milligram equivalents (MME). Includes all opioid medications administered as part of postoperative analgesia, both scheduled and rescue doses. Data will be extracted from electronic medication records and converted using standard MME conversion factors.

SECONDARY OUTCOMES:
Time to First Rescue Opioid Administration | 0-48 hours postoperatively
  Time in hours from the end of surgery to the first administration of rescue opioid analgesia (5 mg intravenous oxycodone) triggered by a Numerical Rating Scale (NRS) pain score ≥ 4 or patient request.
Numerical Rating Scale (NRS) Pain Scores at Rest | 4 hours postoperatively
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Pain will be assessed by blinded study personnel at predefined intervals.
Numerical Rating Scale (NRS) Pain Scores at Rest | 8 hours postoperatively
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Pain will be assessed by blinded study personnel at predefined intervals.
Numerical Rating Scale (NRS) Pain Scores at Rest | 12 hours postoperatively
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Pain will be assessed by blinded study personnel at predefined intervals.
Numerical Rating Scale (NRS) Pain Scores at Rest | 24 hours postoperatively
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Pain will be assessed by blinded study personnel at predefined intervals.
Numerical Rating Scale (NRS) Pain Scores at Rest | 48 hours postoperatively
  Pain intensity at rest measured using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Pain will be assessed by blinded study personnel at predefined intervals.
Numerical Rating Scale (NRS) Pain Scores During Movement | 4 hours postoperatively
  Pain intensity during passive hip flexion or standardized physiotherapy-assisted mobilization using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Assessments performed by blinded study staff.
Numerical Rating Scale (NRS) Pain Scores During Movement | 8 hours postoperatively
  Pain intensity during passive hip flexion or standardized physiotherapy-assisted mobilization using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Assessments performed by blinded study staff.
Numerical Rating Scale (NRS) Pain Scores During Movement | 12 hours postoperatively
  Pain intensity during passive hip flexion or standardized physiotherapy-assisted mobilization using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Assessments performed by blinded study staff.
Numerical Rating Scale (NRS) Pain Scores During Movement | 24 hours postoperatively
  Pain intensity during passive hip flexion or standardized physiotherapy-assisted mobilization using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Assessments performed by blinded study staff.
Numerical Rating Scale (NRS) Pain Scores During Movement | 48 hours postoperatively
  Pain intensity during passive hip flexion or standardized physiotherapy-assisted mobilization using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst pain). Assessments performed by blinded study staff.
Quadriceps Muscle Strength | 4 hours postoperatively
  Motor strength of knee extension and hip adduction assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal strength) by two blinded assessors.
Quadriceps Muscle Strength | 8 hours postoperatively
  Motor strength of knee extension and hip adduction assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal strength) by two blinded assessors.
Quadriceps Muscle Strength | 12 hours postoperatively
  Motor strength of knee extension and hip adduction assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal strength) by two blinded assessors.
Quadriceps Muscle Strength | 24 hours postoperatively
  Motor strength of knee extension and hip adduction assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal strength) by two blinded assessors.
Quadriceps Muscle Strength | 48 hours postoperatively
  Motor strength of knee extension and hip adduction assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal strength) by two blinded assessors.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperatively
  Presence of nausea, vomiting, or use of antiemetic medications documented by nursing staff and confirmed by blinded investigators.
Time to First Mobilization | 0-48 hours postoperatively
  Time in hours from the end of surgery until the patient is able to stand with physiotherapist assistance. Early mobilization follows institutional enhanced recovery protocols.
Adverse Events Related to Regional Anesthesia | Up to 48 hours postoperatively
  Incidence of block-related complications including vascular puncture, local anesthetic systemic toxicity, persistent sensory deficit, motor deficit, or nerve injury as documented in hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznań University of Medicla Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome analyses will be made available to other researchers upon reasonable request. Shared data will include demographic variables, intraoperative information, block-related details, pain scores, opioid consumption, motor assessments, and adverse events. No direct identifiers or protected health information will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will become available 12 months after publication of the primary results and will remain accessible for 5 years.
Access Criteria: Researchers must submit a methodologically sound proposal describing the intended use of the data. Requests will be reviewed by the study investigators. Data will be shared through secure, password-protected transfer methods. A data-sharing agreement will be required before access is granted.